CLINICAL TRIAL: NCT00272220
Title: Longitudinal Randomized Controlled Study of Modified Directly Observed HAART in Mozambique
Brief Title: Longitudinal Study of HAART, Social Networks, & Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mozambique Ministry of Health (Unknown); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-9137-G 01; TAP:HIV-AIDS/MS-DPC/GACOPI/04
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Acquired Immunodeficiency Syndrome; Antiretroviral Therapy, Highly Active; Randomized Controlled Trials; Africa; Adherence; Treatment Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): receive 6-week intervention of peer-delivered mDOT
  Interventions: Behavioral: modified directly observed therapy (mDOT)
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: modified directly observed therapy (mDOT) — Peers individually administered the 6-week mDOT intervention at the Beira Day Clinic to mDOT participants during their morning weekday dose. Evening and weekend doses were not observed. Nighttime and weekend doses were self-administered. As part of the daily interaction with participants, peers provided social support, information about the benefits and side effects of HAART, how to address stigma's effect on adherence, and encouragement to participate in community support groups. The peers also provided an important link between the individual and other members of the HIV clinic team and the community.
  Arms: 1

SUMMARY:
Our study is a randomized controlled trial that aims to evaluate the effectiveness of modified directly observed therapy (mDOT) to (1) increase both short and long term adherence to HAART treatment, and (2) improve clinical outcomes associated with HAART therapy.

Our hypothesis is that modified directly observed therapy (mDOT) during the initial 6 weeks of HAART, supervised primarily by HIV-positive lay activists, will improve adherence and clinical outcomes compared with those that do not have supervised mDOT. We also hypothesize that the benefits of mDOT will be achieved through a variety of mediators that will result from the social interactions the patients will have with the activists. These mediators include improved social support, improved knowledge about HAART, reduced stigma, and improved self-efficacy.

DETAILED DESCRIPTION:
To test this hypothesis, we intend to randomize 350 ARV naïve patients starting HAART to either receive mDOT for the initial 6 weeks of treatment or standard adherence support. Both intervention and control groups will receive standard HIV care that includes HAART medications free of charge, clinical and laboratory follow-up, psychosocial adherence support by a trained social worker, and referral to community-based peer support groups. Patients in the intervention group will in addition to stand care, receive their morning weekday dose of a twice-daily HAART regimen under DOT in clinic for 6 weeks. Nighttime and weekend doses are self-administered. A group of HIV-positive DOT activists, who are trained and paid lay-clinic personnel, will be primarily responsible for the direct observation of treatment in the mDOT group. In addition to observing treatment, DOT activists will provide counseling, education, and emotional support to patients, and will also locate patients not presenting for DOT on the same day. Although the HIV activists may also provide psychosocial and adherence support to specific patients in the control group, this support will only be a daily and formalized part of care in the group randomized to mDOT.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ persons initiating HAART
* Adults and children over the age of 18
* Reside in or around Beira Mozambique
* Willing and able to provide consent to participate

Exclusion Criteria:

* Physically or mental incapable to make daily clinic visits
* Psychotic or demented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2004-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Self-report - 7 & 30 day recall | at 6 months and 12 months

SECONDARY OUTCOMES:
Change in CD4 count | from baseline to 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Pearson, PhD(C), Principal Investigator — University of Washington; Stephen Gloyd, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Beira Day Hosptial - Central Hospital, Beira, Sofala, Mozambique